CLINICAL TRIAL: NCT07215715
Title: Myocardial & Hepatic Shear Wave Velocity Measurements in Patients With Non-Reduced-Ejection Fraction Heart Failure and Control Subjects - US Benchmarking Clinical Study
Brief Title: US Benchmarking Clinical Study
Acronym: EMS-CT-1
Status: Recruiting | Type: Observational
Sponsor: eMyosound SAS (Industry)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: EMS-CT-1
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction; HFmrEF; ATTR-CM (Transthyretin Amyloid Cardiomyopathy); Left Ventricular Hypertrophy; Cardiac Amyloidosis
Keywords: Shear Wave Velocity; non-invasive ultrasound elastography; US Benchmarking Clinical Study; Heart Failure; Cardiac Amyloidosis; ATTR-CM
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Amyloid Neuropathies, Familial; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure with LVEF > 40% and LVH with ATTR-CM: heart failure (HF) with left ventricular ejection fraction (LVEF) > 40% and left ventricular hypertrophy (LVH) with transthyretin amyloidosis with cardiomyopathy (ATTR-CM)
- Heart Failure with LVEF > 40% and LVH, without ATTR-CM: Heart Failure with LVEF > 40% and LVH, without ATTR-CM
- Control group of patients without heart failure or cardiomyopathy: Control group of patients without heart failure or cardiomyopathy.

SUMMARY:
The goal of this observational study is to measure shear wave velocity (SWV) in patients with non-reduced left ventricular ejection fraction (LVEF) heart failure and left ventricular hypertrophy, with or without transthyretin amyloidosis with cardiomyopathy (ATTR-CM), and in control subjects without heart failure or cardiomyopathy.

The main question it aims to answer is:

• Can SWV be used to measure myocardial and liver stiffness in the study's target populations? Researchers will compare patients with ATTR-CM, patients without ATTR-CM, and a control group to determine the distributions of SWV in each population.

Participants will:

* Have a standard cardiology assessment, including a physical exam, blood work, and an echocardiogram.
* Undergo an investigational assessment with the eMyosound LYRA device to measure SWV in their myocardium and liver.
* Have the investigational assessment repeated by a second observer to assess measurement reliability.

DETAILED DESCRIPTION:
This is a multicenter, prospective, consecutive cross-sectional study with three parallel arms and non-competitive enrollment. The study is designed to advance the clinical understanding of myocardial and hepatic stiffness by using a novel ultrasound elastography device, the eMyosound LYRA. The prospective design is essential because this elastographic assessment is not yet part of standard care, and the investigational device is being made available specifically for this research. Consecutive recruitment will be used to minimize selection bias by inviting all eligible patients to participate. The cross-sectional design means that no longitudinal follow-up visits are required, making the study feasible for a single-visit assessment.

The primary objective is to determine the shear wave velocity (SWV) in the left ventricle, right ventricle, and liver of three distinct patient populations as specified in the Groups and Interventions section of this form.

The study also aims to establish the device's proportion of patients in whom SWV can be estimated, to characterize the distribution of various myocardial and hepatic SWV measurements, and to compare these distributions between the three study arms. We will also investigate the statistical associations between SWV and a range of clinical, ECG, laboratory, and echocardiographic variables to better understand how these parameters correlate with myocardial stiffness. A key part of our methodology involves a test-retest procedure with two independent observers to establish the within-observer repeatability and between-observer reliability of the SWV measurements.

Study Conduct and Procedures The study will enroll a total of 150 analyzable participants (50 per arm) from three medical centers. The total enrollment may reach up to 180 to account for potential dropouts or non-contributing data. The study is confined to a single visit for each participant, with a total estimated duration of 2.5 hours.

At the single visit, after informed consent is signed, patients will undergo a series of assessments. A standard medical history and physical examination will be performed. Patients will also receive a 12-lead ECG, blood work (including NT-proBNP and hsTnT), and a standard echocardiogram with a wide range of measurements.

Following these standard cardiology assessments, the investigational elastographic assessment will be performed with the eMyosound LYRA device, a Class II medical device for real-time sonographic imaging, shear wave measurement, and electrocardiographic recording. The assessment includes two types of shear wave measurements using the device's M3-5 LYRA probe:

Myocardial Shear Wave Velocity (SWV): Measurements will be taken in specific myocardial regions of interest (ROIs), including the right ventricular anterior free wall (RVAW), left ventricular anteroseptal wall (LVAW), and interventricular septum (IVS). These measurements are acquired in both parasternal long-axis (PLAX) and parasternal short-axis (PSAX) views, and the IVS is also measured in the apical 4-chamber (A4C) view.

Hepatic Shear Wave Velocity (SWV): The operator will measure SWV in two distinct ROIs of the liver's right lobe.

The types of measurements include Acoustic Radiation Force Induced Shear Waves (ARF-SWV), which are performed during diastasis, and Natural Shear Waves (N-SWV), which are produced by cardiac movements. For the test-retest procedure, each of the two observers will attempt to acquire 20 repeated valid measurements for each target ROI.

Risk and Safety Management The study is designed to minimize risks, which are similar to those of other echocardiographic devices. Risk management is handled by respecting the device's indications and contraindications and providing detailed training and technical support to investigators. The potential benefit to participants is a free, thorough cardiological assessment. A Data and Safety Monitoring Board (DSMB) will provide independent oversight, review all adverse events, and make recommendations to the sponsor.

Statistical Analysis The study is primarily descriptive and exploratory. The target sample size is 150 analyzable patients. The final analysis will be performed once all participants have completed the study. Two interim analyses are planned: a qualitative analysis after the first 15 patients to check for safety issues and a quantitative analysis after the first 75 patients to check data quality.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Common to all three Study Arms:

1. Male or female age ≥ 60 years
2. Signed informed consent and able to comply with protocol

   Inclusion Criteria Common to the Heart Failure with non-reduced left ventricular ejection fraction (LVEF) with or without transthyretin amyloid cardiomyopathy (ATTR-CM) Arms:
3. Patients meeting the Universal Definition of Heart Failure & HeartShare study criteria.
4. LVEF >40% on the last available imaging study
5. Left ventricular hypertrophy (LVH) defined as left ventricular mass index (mass/BSA) in female > 95 g/m², in male > 115 g/m² according to American Society of Echocardiography/European Association of Cariology (ASE/EAC) guidelines42 OR as interventricular septum (IVS) thickness ≥12 mm

   Inclusion criterion specific to HF with non-reduced LVEF without ATTR-CM Arm:
6. Negative (grade 0) Pyrophosphate (PYP) scintigraphy within 24 months prior to the enrolment in the study OR Simple Score <643 OR negative endomyocardial biopsy

   Inclusion criterion specific to HF with non-reduced LVEF with ATTR-CM Arm:
7. ATTR-CM objectively confirmed and classified at any time prior to the enrollment in the study, with monoclonal protein AL amyloidosis ruled out, according to American Heart Association (AHA) 2020 criteria

   Inclusion criteria in Control Subjects:
8. No diagnosis of HF or cardiomyopathy according to the universal definition of Heart Failure
9. No diagnosis of Transthyretin amyloid cardiomyopathy (ATTR-CM) or Amyloid light-chain (AL) amyloidosis

Exclusion Criteria:

Exclusion criteria common to the three arms:

1. Pregnant OR pre-menopausal woman
2. Vulnerable patients
3. Acute Coronary Syndrome within 30 days
4. Heart rate greater than 130 beats/minute at the time of the measurements
5. Atrial fibrillation or flutter at the time of SWV measurement (history of AF is authorized provided they patient is in sinus rhythm at the time of the measurements)
6. Any clinically significant cardiac arrhythmia at the time of SWV measurement
7. Poor echogenicity preventing accurate ultrasound measurements
8. Patients with segmental wall motion abnormalities thought to be due to myocardial infarction.
9. Severe mitral or aortic valve disease (regurgitation or stenosis) excluded if the cause is other than ATTR (e.g., prolapse, endocarditis, prosthetic valve.)
10. Severe tricuspid valve disease (regurgitation or stenosis) excluded if the causes are other than ATTR.
11. Distance from skin to IVS ≥ 8 cm
12. Any prosthetic mechanical valve
13. Patients with mechanical cardiac assist devices other than pacemakers or defibrillators
14. Heart, lung, liver or kidney transplant history or expected in the next year
15. Severe renal impairment with eGFR < 15 mL/min/1.73m² or end-stage renal disease or patient on dialysis.
16. Presence of any competing life-threatening risk over the next 12 months
17. Complicated uncontrolled diabetes mellitus HbA1c ≥9% with target organ damage.
18. Uncontrolled and persistent high-blood pressure with diastolic pressure > 100 mmHg or systolic pressure > 160 mmHg at the time of the measurement.
19. Acute decompensated state such as volume overload, etc. in the opinion of the study investigator
20. Skin abnormalities, infections, or open wounds at the site of the SVW measurement
21. Liver disease, at least moderate

    Exclusion criteria in both the HF with non-reduced LVEF with or without ATTR-CM Arms:
22. Known inherited cardiomyopathy, infiltrative cardiomyopathy (other than ATTR-CM for the study arm for ATTR-CM), cardiomyopathy from muscular dystrophies, cardiomyopathy with reversible causes (e.g., stress cardiomyopathy), hypertrophic cardiomyopathy or known pericardial constriction
23. History of treatment for ATTR-CM with Transthyretin (TTR) depleters

    Exclusion criteria Specific to Control Subjects:
24. Any diagnosis of cardiomyopathy or HF, whatever the cause46
25. LVH based on LV mass index female >95 g/m², in male ≥115 g/m² OR IVS thickness ≥12 mm unless thought to be due to athlete's heart

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of three distinct groups, or cohorts, participating in a multicenter study. The total target enrollment is 150 analyzable patients, with 50 patients per arm from each of the three sites. An additional 30 patients may be enrolled to account for non-contributing data. The study focuses on individuals aged 60 and older, with no upper age limit.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures are the shear wave velocity (SWV) measurements extracted from the eMyosound LYRA device acquisitions. | single study visit of a duration of approximatively 2.5 hours
  These measurements include:
  Myocardial Acoustic Radiation Force (ARF)-SWV, defined as the velocity projected along the muscle fibers during diastasis.
  Myocardial Natural (N)-SWV, measured during both mitral valve closure (MVC) and aortic valve closure (AVC).
  Hepatic ARF-SWV, measured in two distinct regions of the right liver lobe.

SECONDARY OUTCOMES:
The secondary outcome measures are comprehensive and are used to establish distributions, assess device performance, and explore associations with clinical data | single-study visit of a duration of approximatively 2.5 hours
  The proportion of patients for whom SWV can be estimated in each region of interest (ROI) and each view [Parasternal Long Axis (PLAX) view, Parasternal Short Axis (PSAX) view, Apical Four Chamber (A4C) view].
Distribution of myocardial Acoustic Radiation Force - Shear Wave Velocity (ARF-SWV) and myocardial Natural - Shear Wave Velocity (N-SWV). | single-study visit of a duration of approximatively 2.5 hours
  Establish the distribution of myocardial ARF-SWV and myocardial N-SWV.
Distribution of hepatic ARF-SWV. | single-study visit of a duration of approximatively 2.5 hours
  Establish the distribution of hepatic Acoustic Radiation Force - Shear Wave Velocity (ARF-SWV).
Within-observer repeatability of Shear Wave Velocity (SWV) measurements per Region of Interest (ROI) | single-study visit of a duration of approximatively 2.5 hours
  Establish the within-observer repeatability of SWV measurements per ROI
Between-observer reliability of SWV measurements per ROI | single-study visit of a duration of approximatively 2.5 hours
  Establish the between-observer reliability of SWV measurements per ROI
Comparison of SWV distributions between the three study arms | single-study visit of a duration of approximatively 2.5 hours
  Compare the SWV distributions between the three study arms
Statistical associations between the various myocardial and hepatic SWVs and study assessment variables | single-study visit of a duration of approximatively 2.5 hours
  Identify the statistical associations between the various myocardial SWVs and the clinical, electrocardiogram (ECG), laboratory, and echocardiographic variables
Safety of the procedure | single-study visit of a duration of approximatively 2.5 hours
  Establish the safety of the procedure, documented by the number and severity of adverse events during the study visits until discharge
Identify the statistical associations between the various hepatic SWVs and study assessment variables | single-study visit of a duration of approximatively 2.5 hours
  Identify the statistical associations between the various hepatic SWVs and the clinical, electrocardiogram (ECG), laboratory, and echocardiographic variables

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Sarda, Study Director — eMyosound SAS
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No